CLINICAL TRIAL: NCT01647178
Title: The Influence of the TORQ Sternal Closure Assistance Device on Post-Operative Pain, Pulmonary Function and Quality of Life Compared to Traditional Manual Wire Closure: A Randomized Controlled Trial.
Brief Title: TORQ Clinical Study
Acronym: TORQClin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kardium Inc. (Industry)
Collaborators: St. Paul's Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H11-00310
Record Dates: First submitted 2012-07-17; First posted 2012-07-23 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Post Cardiac Surgery; Sternal Closure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual closure (Active Comparator): Patients are closed with a manual, straight wire, conventional closure technique
  Interventions: Procedure: Conventional closure
- TORQ closure (Active Comparator): Patients are undergo a TORQ assisted sternal closure
  Interventions: Procedure: TORQ assisted sternal closure

INTERVENTIONS:
Procedure: TORQ assisted sternal closure
  Other Names: TORQ (Manufacturer: Kardium, Richmond, Canada)
  Arms: TORQ closure
Procedure: Conventional closure
  Other Names: Straight wire closure
  Arms: Manual closure

SUMMARY:
The proposed trial is to evaluate the use of the TORQ closure assistance device and how it affects pain in the sternum, breathing and quality of life compared to traditional use of needle drivers or similar to close sternal wires.

ELIGIBILITY:
Inclusion Criteria:

* Referred for elective cardiac surgery at St Paul's Hospital
* Expected to live greater than 12 months
* Capable of giving written informed consent
* Willing to participate in follow-up
* Greater than 18 years of age, and of legal age of consent in host country

Exclusion Criteria:

* Patient has had previous median sternotomy, requiring redo sternotomy
* Surgeon has, prior to enrollment, elected to use alternative closure technique to the interrupted single wire circlage technique (e.g. Figure of 8 technique)
* Surgeon has elected, prior to enrollment. to treat with the TORQ as a prophylactic measure (e.g. in high risk cases where use of the TORQ has been shown to be effective in preventing dehiscence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Respiratory function | Pre-op, 2 and 4 days Post-op
Pain Score | 2, 4, 14, 30 and 90 days post op
  Patient reported pain on a scale of 1 to 10 for breathing, coughing and walking

CONTACTS AND LOCATIONS:
Overall Officials: James Abel, MD, Principal Investigator — St. Paul's Hospital, Canada
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada